CLINICAL TRIAL: NCT01900600
Title: Substudy of the the CANTOS Trial (Interleukin-1 Blockade With Canakinumab to Improve Exercise Capacity in Patients With Chronic Systolic Heart Failure and Elevated Hs-CRP; CACZ885M2301)
Brief Title: Interleukin-1 Blockade With Canakinumab to Improve Exercise Capacity in Patients With Chronic Systolic Heart Failure and Elevated High Sensitivity C-reactive Protein (Hs-CRP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: HM13782; 20110521 (Other: WIRB)
Record Dates: First submitted 2013-07-06; First posted 2013-07-16 (Estimated); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: Prior Acute Myocardial Infarction; Evidence of Systemic Inflammation (C Reactive Protein Plasma >2 mg/l); Reduced Left Ventricle Ejection Fraction (<50%); Symptoms of Heart Failure (NYHA Class II-III)
MeSH Terms: interventions — Exercise Test; Caves

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Cardiopulmonary exercise test; Other: Echocardiogram
- Canakinumab 50 mg quarterly (Active Comparator): Canakinumab 50 mg quarterly
  Interventions: Other: Cardiopulmonary exercise test; Other: Echocardiogram
- Canakinumab 150 mg quarterly (Active Comparator): Canakinumab 150 mg quarterly
  Interventions: Other: Cardiopulmonary exercise test; Other: Echocardiogram
- Canakinumab 300 mg quarterly (Active Comparator): Canakinumab 300 mg quarterly
  Interventions: Other: Cardiopulmonary exercise test; Other: Echocardiogram

INTERVENTIONS:
Other: Cardiopulmonary exercise test — All patients will undergo a first CPX prior to initiation of treatment, a second one after 3 months, and a third one after 12 months of treatment.
  Other Names: Cardiopulmonary exercise test (CPX)
Other: Echocardiogram — An echocardiogram (ultrasound of the heart) will be performed prior to initiation of treatment and then again 12 months later.
  Other Names: Echocardiogram or Echo

SUMMARY:
The proposed study is a sub-study of the CANTOS trial (A randomized, double-blind, placebo-controlled, event driven trial of quarterly subcutaneous canakinumab in the prevention of recurrent cardiovascular events among stable post-myocardial infarction patients with elevated high sensitivity C-reaction protein (hsCRP) [CACZ885M2301]).

The study proposes to perform serial Cardiopulmonary Exercise Tests (CPX) to prospectively measure changes in aerobic exercise capacity in patients with prior myocardial infarction (MI), elevated C reactive protein plasma levels, and symptomatic heart failure with reduced systolic function, who are enrolled in the main CANTOS trial and are randomly assigned to Canakinumab (3 different doses) or Placebo.

The subjects enrolled in this substudy will undergo repeated CPX and echocardiograms over the first 12 months of the CANTOS trial. The subjects will received the experimental treatment as randomized in the main CANTOS trial and they will not receive any additional experimental treatment as part of the sub-study.

This study is a an Investigator-initiated (Dr. Abbate) single-center (Virginia Commonwealth University) sub-study of the CANTOS trial, supported by Novartis pharmaceuticals.

DETAILED DESCRIPTION:
Patients enrolled in the CANTOS trial (with prior acute myocardial infarction [>30 days] and elevated C reactive protein levels [CRP>2mg/l]) who also have reduced left ventricular ejection fraction (LVEF<50%) and are symptomatic for heart failure (New York Heart Association symptoms class II-III) will be offered to take part in this sub-study at the Virginia Commonwealth University site.

As part of the sub-study, patients will undergo a cardiopulmonary exercise test (CPX) at baseline prior to initiation of treatment, then repeated at 3 and 12 months, and a transthoracic echocardiogram at baseline and at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* all criteria listed in the CANTOS trial (CACZ885M2301)
* left ventricular ejection fraction <50%
* symptoms of heart failure (NYHA class II-III)

Exclusion Criteria:

* all criteria listed in the CANTOS trial (CACZ885M2301)
* inability to complete a treadmill exercise test
* conditions preventing interpretation of the cardiopulmonary test (arrhythmias, ischemia, hypertension, pulmonary disease)

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-04; Primary Completion 2015-01-08 (Actual); Study Completion 2015-01-08 (Actual)

PRIMARY OUTCOMES:
Peak oxygen consumption (VO2) | 3 months
  Difference in the interval change from baseline in peak VO2 at 3 months following a single dose of CANAKINUMAB 50 mg subcutaneous, 150 mg subcutaneous, or CANAKINUMAB 300 mg subcutaneous [all three groups combined] when compared with the interval change in placebo (placebo-corrected interval change).

SECONDARY OUTCOMES:
Peak VO2 change | 12 months
  Difference in the interval changes from baseline and 12 months in peak VO2 comparing CANAKINUMAB (all doses) with placebo
Ventilatory efficiency (VE/VCO2 slope) change | 12 months
  Difference in the interval changes from baseline and 3 months in the VE/VCO2 slope comparing CANAKINUMAB (all doses) with placebo
OUES | 12 months
  Difference in the interval changes from baseline and 12 months in oxygen utilization efficiency slope (OUES) comparing CANAKINUMAB (all doses) with placebo
LVEF change | 12 months
  Difference in the interval changes from baseline and 12 months in left ventricular ejection fraction (LVEF) comparing CANAKINUMAB (all doses) with placebo
Diastolic function change | 12 months
  Difference in the interval changes from baseline and 12 months in E/E' (diastolic function) comparing CANAKINUMAB (all doses) with placebo

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Abbate, MD, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

REFERENCES:
- [Background] Ridker PM, Thuren T, Zalewski A, Libby P. Interleukin-1beta inhibition and the prevention of recurrent cardiovascular events: rationale and design of the Canakinumab Anti-inflammatory Thrombosis Outcomes Study (CANTOS). Am Heart J. 2011 Oct;162(4):597-605. doi: 10.1016/j.ahj.2011.06.012. Epub 2011 Sep 14. PMID 21982649
- [Background] Abbate A, Van Tassell BW, Biondi-Zoccai GG. Blocking interleukin-1 as a novel therapeutic strategy for secondary prevention of cardiovascular events. BioDrugs. 2012 Aug 1;26(4):217-33. doi: 10.1007/BF03261881. PMID 22571369
- [Derived] Trankle CR, Canada JM, Cei L, Abouzaki N, Oddi-Erdle C, Kadariya D, Christopher S, Viscusi M, Del Buono M, Kontos MC, Arena R, Van Tassell B, Abbate A. Usefulness of Canakinumab to Improve Exercise Capacity in Patients With Long-Term Systolic Heart Failure and Elevated C-Reactive Protein. Am J Cardiol. 2018 Oct 15;122(8):1366-1370. doi: 10.1016/j.amjcard.2018.07.002. Epub 2018 Jul 20. PMID 30244844
- See also: Main CANTOS website — http://www.thecantos.org/cantos-summary.html